CLINICAL TRIAL: NCT00994032
Title: Analysis of the Impact in the Quality of Life of Patients With Pain Secondary to Osteoporotic Vertebral Fractures Receiving Conservative Treatment Versus Percutaneous Vertebroplasty
Brief Title: Quality of Life After Vertebroplasty Versus Conservative Treatment in Patients With Painful Osteoporotic Vertebral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Sociedad Española de Radiologia Medica (Unknown)
Responsible Party: Principal Investigator, JORDI BLASCO ANDALUZ, MD, PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCPB-VP
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Spinal Fracture; Osteoporosis; Back Pain
Keywords: vertebroplasty; disability evaluation; outcome assessment; pain measurement
MeSH Terms: conditions — Spinal Fractures; Osteoporosis; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- vertebroplasty (Active Comparator)
  Interventions: Procedure: percutaneous injection of cement into the vertebral body
- Medical Treatment (Active Comparator)
  Interventions: Other: Medical treatment

INTERVENTIONS:
Procedure: percutaneous injection of cement into the vertebral body — percutaneous injection of cement into the vertebral body
  Arms: vertebroplasty
Other: Medical treatment — standard antalgic medical treatment
  Arms: Medical Treatment

SUMMARY:
The purpose of this study is to determine whether percutaneous vertebroplasty is able to improve long-term quality of life in patients with pain secondary to osteoporotic vertebral fractures, compared to conventional medical treatment.

DETAILED DESCRIPTION:
Osteoporotic vertebral fractures are associated with pain and severe disability in a high percentage of patients. Vertebroplasty has become the treatment of choice to alleviate pain in those patients who have not responded to medical treatment.Although several case series and non-randomized studies have shown the effectiveness of vertebroplasty in alleviating pain secondary to osteoporotic vertebral fractures, the long-term effect of this treatment has not been compared to standard medical treatment in a randomized study.

In our study we have analyzed the long-term effect of vertebroplasty in terms of quality of life in patients with painful osteoporotic vertebral fractures, randomizing them into two arms: percutaneous vertebroplasty or conventional medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Painful (pain intensity of at least 4 on a scale from 0 to 10) osteoporotic vertebral fracture between levels T4 and L5
* Fragility; i.e. fracture not in relation with significant trauma
* Recent fracture, pain beginning not earlier than 1 year before inclusion

Exclusion Criteria:

* No vertebral edema on STIR MR images
* Uncorrectable bleeding diatheses
* Active infection
* Substantial retropulsion of bony fragments
* Non-osteoporotic fracture
* Concomitant neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-03; Primary Completion 2011-06-01 (Actual); Study Completion 2011-06-01 (Actual)

PRIMARY OUTCOMES:
Impact into quality of life with the Qualeffo-41 test | Baseline, 2 weeks, 2 months, 6 months and 1 year

SECONDARY OUTCOMES:
Analyze pain alleviation with the Analog Visual Scale | Baseline, 2 weeks, 2 months, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Blasco, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Blasco J, Martinez-Ferrer A, Macho J, San Roman L, Pomes J, Carrasco J, Monegal A, Guanabens N, Peris P. Effect of vertebroplasty on pain relief, quality of life, and the incidence of new vertebral fractures: a 12-month randomized follow-up, controlled trial. J Bone Miner Res. 2012 May;27(5):1159-66. doi: 10.1002/jbmr.1564. PMID 22513649
- See also: International Osteoporosis Foundation — http://www.iofbonehealth.org/